CLINICAL TRIAL: NCT06340152
Title: Multi-Omics for Maternal Health After Preeclampsia
Acronym: MOM-Health
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Louise Laurent, MD/PhD, Professor, University of California, San Diego
Other Study IDs: 808385; U01HG013189-01 (NIH)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Pre-Eclampsia; Pregnancy Induced Hypertension
Keywords: hypertension; pregnancy; pre-eclampsia; postpartum
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low-risk pregnancy: Pregnant subjects with none of the following: chronic hypertension, pregestational diabetes, renal disease, autoimmune disease, history of preterm preeclampsia in a prior pregnancy
- High-risk pregnancy: Pregnant subjects with one or more of the following: chronic hypertension, pregestational diabetes, renal disease, autoimmune disease, history of preterm preeclampsia in a prior pregnancy

SUMMARY:
To develop strategies to identify postpartum women at risk for adverse cardiovascular outcomes and provide them with preventative therapies.

DETAILED DESCRIPTION:
The investigators will recruit and retain a diverse population of pregnant women who are high- and low-risk for hypertensive disorders of pregnancy/preeclampsia (HDP/PE) for longitudinal collection of phenotypic and environmental exposure measures and biosamples for integrative analysis of phenotypic, environmental, and multi-omic data to understand links between development of HDP/PE and associated fetal pathologies during pregnancy, as well as postpartum maternal health. Participation in the study will begin no later than the second trimester of pregnancy (enrollment by 24 weeks of gestation) and continue through the first year postpartum. Over the course of the study, biospecimens and relevant surveys and cardiovascular assessments will be collected at specified intervals/time-points, as outlined in the table below. In-person study visits should take no more than 30 minutes. Relevant medical information collected as part of routine clinical care will be obtained from the electronic medical record (EMR). The study will take place at UCSD and VUMC prenatal clinics and hospital labor and delivery units, or another private location of the participants choosing, such as their home or office.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years of age to 50 years of age
* 10-24 weeks gestation at time of enrollment
* Singleton pregnancy
* Planning to deliver at a study site (UCSD or VUMC)

Exclusion Criteria:

* Inability to give informed consent
* Intrauterine fetal demise
* Fetal genetic or structural anomaly
* Institutionalization for psychiatric disorder, mental deficiency or incarcerated
* Active or history of malignancy requiring major surgery or systemic chemotherapy
* Multi-fetal gestation or a twin demise at any gestational age
* Known maternal or fetal chromosomal anomalies
* Patients who plan to keep their placenta after delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The present research study focuses on hypertensive disorders of pregnancy, thus, it is necessary that pregnant participants be enrolled. Within this population, we aim to enroll at least 200 high-risk and 550 low-risk participants.
  Participation in the study will be limited to individuals who speak either English or Spanish, as study staff members are capable of communication with these individuals, and these languages represent the majority of patients seen at both study sites.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia | 2nd trimester - 13 months postpartum
Gestational hypertension | 2nd trimester - Delivery
Postpartum hypertension | Delivery - 13 months postpartum

SECONDARY OUTCOMES:
Postpartum cardiovascular disease | Delivery - 13 months postpartum

OTHER OUTCOMES:
Other cardiovascular disease | 1st trimester - 13 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Louise Laurent, MD, PhD, Principal Investigator — UCSD; Marni Jacobs, PhD, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes